CLINICAL TRIAL: NCT04881396
Title: Response of Haemodialysis Patients to BNT162b2 mRNA Cov-19 Vaccine
Acronym: ROMANOV
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0125; 2021-A00325-36 (Other: ID-RCB)
Record Dates: First submitted 2021-05-04; First posted 2021-05-11 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Vaccines; Hemodialysis Complication
Keywords: immunogenicity; haemodialysis patients; SARS-Cov2 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All haemodialysed patients with a medical prescription of BTN162b2 mRNA Cov-19 vaccine: Serological response is defined by a 4 fold increase of IgG anti-spike protein of SARS-Cov2 between Day 0 (before vaccination) and after complete vaccination (evaluated at Day 7 - 14 post-boost).
  Interventions: Biological: Evaluation of the immunogenicity of the vaccine in haemodialysis patients

INTERVENTIONS:
Biological: Evaluation of the immunogenicity of the vaccine in haemodialysis patients — The immunogenicity of the vaccine will be evaluated at the peak of vaccine response (Day 7 - Day 14 after the second dose) and 6 and 12 months post vaccination, by the evaluation of humoral IgG anti-spike protein response (seroconversion rate, absolute antibody titers, affinity of antibody) and cellular anti SARS-Cov2 response (number, activation capacity, production of interferon gamma of CD4 and CD8 anti sars cov2 specific T cells)

SUMMARY:
Vaccination against SARS-Cov2 is a necessity for haemodialysis patients because difficulties to maintain a self-isolation (leading to a higher contamination than general population) and an increase of mortality in case of contamination (more than 20% of mortality in this population). However, vaccine efficiency is known to be decreased in haemodialysis patients. This lead critical the rapid description of immunogenicity of anti SARS-Cov2 vaccine in haemodialysis patients.

The aim of this study is to describe the immunogenicity of the BTN162b2 SARS-Cov2 vaccine in haemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Medical prescription of BTN162b2 mRNA Cov-19 vaccine
* Treatment by chronic (>1 month) haemodialysis

Exclusion Criteria:

* Non-recommended vaccination scheme
* Refusal to consent

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by chronic haemodialysis, with initiation of a vaccination by BTN162b2 mRNA Cov-19 with classical scheme
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate after vaccination with BTN162b2 mRNA cov-19 vaccine | The seroconversion rate is evaluated at Day 7-Day 14 after the second dose.
  IgG anti SARS-Cov2 spike protein will be evaluated by ELISA at Day 0 (at the initiation of vaccination) anti Day 7 - Day 14 after the second dose (peak of response).
  The seroconversion is defined by an 4 fold increase of IgG anti SARS-Cov2 spike protein titer between Day 0 and Day 7 - Day 14 after second dose.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Department of Nephrology, Hopital Edouard Herriot, Lyon
  - Department of Nephrology, Centre Hospitalier Lyon Sud, Pierre-Bénite